CLINICAL TRIAL: NCT06567704
Title: Cancer-related Fatigue During Maintenance Immunotherapy for Non-small Cell Lung Cancer (NSCLC): a Qualitative Study
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00116521; ONC-LUN-2401 (Other: Atrium Health)
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Cancer related fatigue; Immune checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-small cell lung cancer (NSCLC): Non-small cell lung cancer (NSCLC) patients treated with with immune checkpoint inhibitor.
  Interventions: Behavioral: Interviews

INTERVENTIONS:
Behavioral: Interviews — Interviews

SUMMARY:
The purpose of this research is to understand cancer related fatigue in patients with non-small cell lung cancer (NSCLC), who are being treated with an immune checkpoint inhibitor.

DETAILED DESCRIPTION:
This is an observational pilot study. The target population includes adult patients diagnosed with NSCLC receiving an immune checkpoint inhibitor and reporting concerns of fatigue to their provider. This study will be conducted at Levine Cancer Institute (LCI) and Atrium Health Wake Forest Baptist Comprehensive Cancer Center (AHWFBCCC). This study consists of qualitative interviews at two-time points, the primary, and the follow-up. During the primary interview, patients with NSCLC will be asked to complete the PROMIS® Fatigue-Short Form 7a consisting of seven items. During the follow-up interviews, participants will be asked about any change in their fatigue and views on physical activity.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of consent.
* Must be able to speak, read, and understand English.
* Participants diagnosed with NSCLC, and:

  * have advanced/metastatic disease who are currently receiving immunotherapy monotherapy, or
  * have locally advanced disease who are currently receiving immunotherapy monotherapy after completing thoracic radiation therapy, or
  * who underwent resection and are currently receiving immunotherapy monotherapy after completing all other perioperative treatment
* Immunotherapy planned to continue for at least three months after the time of study enrollment (to ensure participant remains on IO long enough to obtain study assessments)
* Have completed at least two cycles of immunotherapy.
* Self-reported cancer-related fatigued that impacts daily function.

Exclusion Criteria:

* Participants who have received a dose of chemotherapy (including maintenance pemetrexed) within the past 3 months
* Participants who have received radiation therapy within the past 3 months. Note: a short course of palliative radiation therapy within up to 20 Gy and up to 5 fractions is permissible.
* Diagnosis of dementia.
* Anemia Hgb <10 g/dL.
* Sarcopenia which is being pharmacologically treated with a prescribed appetite stimulant (e.g., megestrol).
* Untreated hypothyroidism.
* Symptomatic heart failure.
* Oxygen dependent lung disease.
* Cognitively unable to complete interviews per investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with non-small cell lung cancer (NSCLC) receiving an immune checkpoint inhibitor and reporting concerns of fatigue to their provider.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Themes from qualitative interviews with patients | At 3 months
  Two semi-structured qualitative interviews will be conducted with 20 patients. Themes will be determined through inductive analysis and will focus on key aspects of symptomatic fatigue, including but not limited to the frequency, duration, and severity of CRF and resulting functional impairments. In addition, history of physical activity before diagnosis, preferences for physical activity to treat CRF, and support needed to adhere to physical activity regimens will be considered. Themes from the first and second interviews will be synthesized to capture changes in fatigue and views on physical activity.

SECONDARY OUTCOMES:
Severity and impact of cancer-related fatigue (CRF) | At 3 months
  The severity of CRF and its impact on day-to-day function will be measured using the PROMIS® Fatigue-Short Form 7a (F-SF) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Dori Beeler, PhD, Principal Investigator — Atrium Health Levine Cancer
Locations (2):
- United States (2):
  - Atrium Health Levine Cancer, Charlotte, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No